

## FUNDAÇÃO UNIVERSIDADE DO ESTADO DE SANTA CATARINA THE RECTOR'S OFFICE – GR

Ethics Committee on Research Involving Human Beings - CEPSH / UDESC

## FREE AND EXCLUDED CONSENT TERM

You are being invited to participate in a research entitled "Effect of preoperative guidance and repercussion in gait after total knee arthroplasty", whose general objective is to evaluate the effect of the presence and absence of guidance / Information delivered prior to surgery in the way you walk and at the level of fear of moving. This project was approved by the Research Ethics Committee of UDESC under number 2,009,097, on April 10, 2017.

For this, you will initially undergo a physical evaluation where tests will be performed to assess your functional capacity, how you walk, and specific questionnaires to assess your symptoms. Each step will always be performed by the same evaluator. After the initial physical evaluation, a lottery will be conducted, and you will be directed to one of the following groups: (1) Group that will receive verbal guidance and a leaflet with information related to their physical condition as well as signs and symptoms in the period after surgery; (2) Group that will receive only verbal guidance. It is worth remembering that this draw will be carried out to guarantee the quality of the study and to discuss which protocol was better in the care to the patients.

The evaluation of the way of walking will be done in the Biomechanics Laboratory of CEFID / UDESC, in three moments: before performing the joint replacement surgery, 6 (six) weeks and 6 (six) months after the surgery. In this assessment you will respond to questionnaires and use four computerized equipment to assess your ability to walk, your ability to sit and stand up from a chair, your muscles' function, and your balance. You should be wearing bathing suits, and measurements of weight and height will be made. Afterwards, reflective markers and electrodes will be attached to the skin with adhesive tape. They are spherical plastic markers that will help our computers perform imaging, and electrodes that only receive electrical information from their muscles. From this

preparation you will be asked to walk barefoot straight on a straight surface for 5 meters for four times, totaling 20 meters. Next it will be marked the time it takes you to get up from a chair, walk for 3 (three) meters, perform a turn, continue walking and sit again. Finally, the reflective electrodes and markers will be removed and you will be asked to climb on a platform to perform posture control tests.

His participation in this research is voluntary and will consist of questions that should be answered without interference or questioning by the researcher and biomechanical evaluation. These procedures pose average risks as they can cause fatigue or increased pain, but will not aggravate your symptoms. You can request intervals or interruptions of the tests at any time during the evaluation. If there is any occurrence during the tests, there will be a physiotherapist qualified for the first visits and in case of need the patient will be referred to the necessary care. Your participation is not mandatory.

Your participation is important so that the multidisciplinary team can work better on the recovery of people who perform knee arthroplasty, including you.

I hereby inform you that you are guaranteed access, at any stage of the study, to any clarification of any doubts. You may, if you need to, contact the Ethics Committee on Research in Human Beings (CEPSH / UDESC) of the State University of Santa Catarina at the following address: Av. Madre Benvenuta, 2007 - Itacorubi - 88.035-001 - Florianópolis - SC, or by phone (48) 3321-8000. You are also guaranteed the freedom to withdraw consent at any time and fail to participate in the study without any harm. I guarantee that the information obtained will be analyzed together with other patients, and no identification of any of the participants will be disclosed. You have the right to be kept up-to-date on the partial results of the surveys and, if requested, we will give you all the information you request. There will be no personal expenses or compensation for the participant at any stage of the study, including examinations and consultations. If there is any additional expense, it will be absorbed by the research budget.

While agreeing to participate in this survey, you may withdraw at any time, including for no reason, by informing the researcher's decision to give up the researcher at the address or telephone numbers below. Even if it is a voluntary participation and of no financial interest, you will not be entitled to any remuneration.

We request your authorization for the use of your data for the production of technical and scientific articles. Your privacy will be maintained by not identifying your name.

Thank you for your participation.

NAME OF RESEARCHER: Bibiana Melher Pereira

TELEPHONE NUMBER: (48) 33218636

ADDRESS: LAPEQ - Posture and Balance Research Laboratory - UDESC / CEFID / Rua Paschoal

Simone, 358, Coqueiros - Florianópolis (SC)

Ethics Committee on Research Involving Human Beings - CEPSH / UDESC

Av. Madre Benvenuta, 2007 - Itacorubi - Phone: (48) 3321-8195

Florianópolis - SC 88035-001

## SIGNATURE OF RESPONSIBLE RESEARCHER\_

## **TERMS OF CONSENT**

I declare that I have been informed of all the investigation procedures and that I have received in a clear and objective manner all the explanations pertinent to the project and that all information about me will be confidential. I understand that in this study, the measurements of the experiments / treatment procedures will be done on me, and that I have been informed that I can withdraw from the study at any time.

| Full name | |
|-----------|--------|
| Signature | |
| Local: | Date:/ |